CLINICAL TRIAL: NCT00812682
Title: Physician and Patient Perception of Adjustable Maintenance Dosing of Symbicort Turbuhaler
Acronym: REALITY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Panagiotis Pontikis, MD, Medical & Regulatory Affairs Director, AstraZeneca Greece, AstraZeneca S.A., Greece
Other Study IDs: D5890L00021
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Perception of Physicians & Patients of AMD
Keywords: SYMBICORT AMD
MeSH Terms: interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Symbicort

SUMMARY:
This study will evaluate the perception of the physicians and the patients about the approved adjustable dosing of Symbicort® 160/4,5. Symbicort maintenance dose will be adjusted up and down within the approved dose range of 1x2 - 4x2 inhalations per day, to the level of asthma symptoms. Patients and physicians perception of this new dosing schedule will be evaluated by means of questionnaires completion and direct questioning.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 6 months history of asthma and treatment with an inhaled corticosteroids for at least 3 months prior to visit 1 and/or a history of short term variation in airway function and asthma symptoms responding promptly to convent
* Patients where use of a combination (inhaled corticosteroid and long acting beta2-agonist is appropriate, i.e. not controlled on inhaled corticosteroids alone).

Exclusion Criteria:

* Asthma exacerbation requiring oral corticosteroid treatment in the four weeks prior to visit 1
* Upper Respiratory Tract Infection in the previous four weeks
* Severe cardiovascular disease or other significant concomitant disease, which may interfere with the conduct of the study.
* Women enrolled in the trial should not be planning pregnancy and should be taking adequate contraceptive measures where appropriate.
* Previous enrollment in a clinical study
* Known or suspected hypersensitivity to budesonide, formoterol or inhaled lactose

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2006-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with the adjustable maintenance dosing schedule | Throughout the study
Physicians' satisfaction with the adjustable maintenance dosing schedule | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, MD, Study Director — Medical & Regulatory Affairs Director, AstraZeneca Greece: 4